CLINICAL TRIAL: NCT04380168
Title: Comparing Effect of Adding Ketamine Versus Dexmedetomidine to Bupivacaine in Pec 11 Modified Block on Postoperative Pain Control in Patients Undergoing Breast Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amira Fathy Hefni,MD-EDIC, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FMASU R 24/2019
Record Dates: First submitted 2020-05-06; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: More Effective Postoperative Analgesia After Modified Radical Mastectomy With Better Drug Combination; More Prolonged Duration of Postoperative Analgesia After Modified Radical Mastectomy With Better Drug Combination

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Modified pec 11 trunk block using ketamine additive (Active Comparator): Ultasound guided modified pec 11 trunk block using ketamie hydrochoride 1mg/kg in 2ml volume added to 30ml bupivacaine 0.25% for trunk analgesia
  Interventions: Procedure: Modified pec11 trunk block
- Modified pec 11trunk block using dexmedetomidine additive (Active Comparator): Ultasound guided modified pec 11 trunk block using dexmedetomidine 1ug/kg in 2ml volume added to 30ml bupivacaine 0.25%
  Interventions: Procedure: Modified pec11 trunk block
- Modified pec 11trunk block without additive (Active Comparator): Ultasound guided modified pec 11 trunk block using bupivacaine 0.25% added to 2ml saline
  Interventions: Procedure: Modified pec11 trunk block

INTERVENTIONS:
Procedure: Modified pec11 trunk block — Ultrasound guided modified pec 11 block injecting local anesthetic with or without adjuvant between pectoralis minor and serratus anterior muscles

SUMMARY:
in our study we are trying to reach to the preferred adjuvant from either ketamine or dexmedetomidine to be added to bupivacaine local anesthetic during pec 11 modified block as regard its efficacy and duration of postoperative analgesia it can maintain after modified radical mastectomy surgery so as to achieve better control of postoperative pain than using local anesthetic alone.

DETAILED DESCRIPTION:
* Type of Study: Randomized controlled trials
* Study Setting: Operating theater of Ain Shams University Hospitals, Cairo, Egypt
* Study Period: 6 months .
* Sampling Method:

Patients will be subdivided randomly into 3 groups :

Group (PC): will receive 30 ml of 0.25%bupivacaine plus 2ml normal saline. Group (PK): will receive 30 ml of 0.25% bupivacaine added to ketamine hydrochloride

1mg/kg diluted in 2ml normal saline. Group(PD): will receive 30 ml of 0.25%bupivacaine added to dexmedetomidine 1ug/kg diluted in 2 ml normal saline. Study Procedure Following local university ethical committee approval, informed consent will be obtained. Details of the anesthetic technique and the study protocol will be fully explained at the preoperative visit, and written consent will be obtained from each patient before inclusion in the study.

In the pre-induction room the patients will be taught how to assess their own pain score using the numerical rating scale (NRS) (0-10; 0 = no pain, 10 = worst imaginable pain) and how to use the device for a patient-controlled analgesia (PCA) .Patients in all groups will receive 5mg oral midazolam ,2 hours prior to surgery.A20 gauge IV cannula will be inserted in the upper limb contralateral to the side of surgery upon reaching the operating room .Before induction of anesthesia electrocardiography (ECG), non-invasive blood pressure (NIBP), arterial oxygen saturation (Sao2), and end-tidal carbon dioxide (EtCo2) will connected to the patient. In all groups general anaesthesia will be induced using 2 μg/kg fentanyl, 2.5mg/kg propofol and 1 mg/kg lidocaine. Endotracheal intubation will be facilitated by 0.5 atracurium and was maintained by 1 MAC sevoflurane in 50% Oxygen /air mixture, and ventilator parameters will be adjusted to maintain normocapnia. The Pecs11 Modified block will be done using in plane approach, an 80 mm needle using linear array ultrasound probe of high frequency (12Hz).

The modified Pec 11 block will be done using two needle approach, an 80 mm needle(PajunkR SonoPlex Stim cannula U.S.A) with the aid of linear array ultrasound probe of high frequency (SonositeR, Inc. U.S.A). The modified Pec 11 block technique: The ultrasound probe will be angled inferolateral from the midclavicular level sagittal plane (same as in infraclavicular brachial plexus block) the axillary artery and veins are located ,then the probe will be moved laterally until the pectoralis minor and serratus anterior muscles are seen, after locating 2nd rib immediately under the axillary artery then the ultrasound probe will move caudally from this position until both the third and fourth ribs are seen , the probe is rotated 90 degrees so that it lies transversally and will move laterally toward the anterior axillary line keeping the third rib at the center so that the lateral border of pectoralis minor is will be identified and at the top of the third rib the serratus anterior muscle will be seen deeper to the pectoralis minor ,the needle then will be advanced from the medial to lateral side parallel to the ultrasound beam and 32ml of the solution will be injected between the pectoralis minor and serratus anterior muscles (8,9).

For each group, the 32ml solution constituents are different, for PC group (the control group) the 32ml solution contain only 0.25% bupivacaine while for group PK it contains 1mg/kg ketamine hydrochloride in addition to bupivacaine ,while for group PD it contains 1ug/kg dexmetomedine in addition to bupivacaine. Surgery started 30 minutes after the block has been given. Fentanyl 0.5ug was given as a bolus if HR or BP rose 20% above the baseline values, Bradycardia (HR<50/minute) is treated with atropine 0.5mg bolus, and hypotension (20% below the baseline values) is treated with 10mg boluses of ephedrine. Patients were extubated after adequate neuromuscular reversal using atropine 0.02mg/kg and 0.05mg/kg neostigmine.

After that the patients were transferred to post-anaesthesia care unit where they were followed up and assessed for the following parameters: O2 saturation(spo2),Respiratory rate(RR), Non-invasive blood pressure(NIBP),Heart rate(HR), and Sedation agitation scores using Richmond Agitation Sedation Scale(RASS)( +4=combative +3=very agitated +2=agitated +1=restless 0=alert and calm,-1=drowsy,-2=light sedation,-3=moderate sedation ,-4=deepsedation,-5=unarousable sedation) (11) will be measured 5, 10, 20, 30, 45, and 60 min postoperatively . Episodes of postoperative nausea and vomiting, sedation scale above 2,any psychological complications (as hallucinations, dreams),are recorded and treated. nausea and vomiting will be treated by ondansetron 4mg IV, if sedation scale scores< -2 patient will receive flumazenil 0.15mg IV over 15secnds ,and if patient manifest hallucination or RASS >+1, 1mg Midazolam IV will be given.

Pain scores(NRS) at rest and movement of ipsilateral arm will be recorded every hour for 24 hour postoperatively .Total intraoperative fentanyl consumption ,and total postoperative morphine consumption for the first 24 hours postoperative will be calculated and the time of the first request of analgesic will be recorded. When analgesia is requested postoperatively( once the pain is expressed by the patient or the NRS was>3 ) an initial morphine bolus of 0.1mg/kg followed by 1mg bolus with a lockout periods of 15 minutes with no background infusion allowed. At the end of 24 h, the patient's satisfaction about the post-operative analgesia which was rated on a three-point scale, i.e., good = most satisfied, average = somewhat satisfied, poor= dissatisfied, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ASA1,11,111 between 18 and 60 years scheduled for modified radical mastectomy

Exclusion Criteria:

* Patients with history of advanced cardiac disease
* Patients having sepsis,
* Patients with prior surgery in areas above or below the clavicle or in the axillary region,
* Patients with opioid dependence or alcohol or drug abuse,
* Patients with coagulopathy
* Patients with psychiatric illness that prevent them from proper perception and assessment of pain.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 5 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Total postoperative morphine consumption over the first 24 hours postoperative | "through study completion ,an average of one year"
  number value
The time to first request of analgesic postoperatively | "through study completion ,an average of one year"
  time

SECONDARY OUTCOMES:
pain scores at rest and active movement of ipsilateral arm | "through study completion ,an average of one year"
  number value
intraoperative fentanyl requirements | "through study completion ,an average of one year"
  number value

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university Hospitals, Cairo, Egypt